CLINICAL TRIAL: NCT03925103
Title: Ergonomical Assessment of Three-Dimensional Versus Two-Dimensional Thoracoscopic Lobectomy for Lung Cancer
Brief Title: Assessment of Ergonomics in 3D vs 2D Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Eugenio Pompeo, Principal Investigator, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-1RT
Record Dates: First submitted 2019-02-27; First posted 2019-04-23 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Early Stage Non-small-cell Lung Cancer (Stage 1-2)
Keywords: VATS; Lobectomy; 3D VATS; VATS Ergonomics; Non small cell lung cancer; Three-dimensional thoracoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: One to one parallel assignment to each treatment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D VATS lobectomy (Experimental): Patients undergo thoracoscopic lobectomy by a three-dimensional display system
  Interventions: Procedure: 3D VATS lobectomy
- 2D VATS lobectomy (Active Comparator): Patients undergo thoracoscopic lobectomy by a two-dimensional display system
  Interventions: Procedure: 2D VATS lobectomy

INTERVENTIONS:
Procedure: 3D VATS lobectomy — pulmonary lobectomy carried out by video-assisted thoracoscopic surgery with a 3 dimensional display system
  Arms: 3D VATS lobectomy
Procedure: 2D VATS lobectomy — pulmonary lobectomy carried out by video-assisted thoracoscopic surgery with a 2 dimensional display system
  Arms: 2D VATS lobectomy

SUMMARY:
Video-assisted thoracic surgery (VATS) pulmonary lobectomy is currently widely employed as the first treatment option for surgical management of early stage (stage I-II) non-small-cell-lung-cancer (NSCLC).

Thanks to recent technological advances in high definition display systems, three dimensional VATS (3D) has been developed in an attempt of overcoming some optical limits of two dimensional (2D) VATS.

In this single center randomized trial our aim is to comparatively assess ergonomics of 3D versus 2D VATS lobectomy for early stage NSCLC.

DETAILED DESCRIPTION:
Video-assisted thoracic surgery (VATS) is widely employed for pulmonary lobectomy in early stage non-small-cell-lung-cancer (NSCLC). Indeed, VATS is thought to represent an optimal minimally invasive surgical option which is deemed superior to conventional thoracotomy since it enables smaller incisions with no rib spreading thus minimizing both postoperative pain and hospital stay.

For over than three decades, several thoracic surgeons adopted VATS for anatomical lung resection using two-dimensional (2D) display systems. However, a 2D image lacks depth of perception which may negatively affect surgical manoeuvring.

Three dimensional (3D) display systems for VATS can offer superior magnified vision of the surgical field and better perception of depth during surgical manoeuvring potentially shortening learning curve, which may thus overcome some optical limitations of 2D systems.

In this single center randomized trial our aim is to comparatively assess ergonomics of 3D versus 2D VATS lobectomy for early stage (stage I-II) NSCLC. For this purpose we compared three ergonomical domains: exposure, instrumentation and maneuvering with the aid of a scoring scale entailing analysis of 5 main technical steps: vein, artery bronchus, lymph node and fissure score.

The evaluation process of the five surgical steps was carried out by 4 thoracic surgeons who individually scored all recorded operations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical NSCLC early stage (stage I-II).
* Both forced expiratory volume in one second (FEV1) and diffusion capacity of carbon monoxide (DLCO)>60%
* Both predicted postoperative (PPO) FEV1 and PPO DLCO >35%
* American Society of Anesthesia (ASA) score<=2
* Body mass index (BMI) >18 <28

Exclusion Criteria:

* Clinical NSCLC stage> II
* History of Neoadjuvant chemotherapy or radiotherapy
* Radiologic evidence of extensive pleural adhesions.
* Age <18 or >80 years.
* Patients with previous pleurodesis or thoracotomy in the affected hemithorax.
* Patients who will undergo surgical lung resection other than lobectomy.
* Patients with severe comorbidity contraindicating lobectomy.
* Patients refusal or noncompliance to general surgery and one-lung ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
a difference ≥10% in the score calculated for the maneuvring ergonomical domain. | one week after surgery
  3 ergonomical domains: exposure, instrumentation and maneuvering are assessed by 4 thoracic surgeons using a new scoring scale (score range 1, unsatisfactory to 3 excellent). Primary outcome is a difference ≥10% (sd=0.3) in at least one of the evaluated domains.

SECONDARY OUTCOMES:
Operative time | during surgery
  Total duration (min) of the surgical procedure from first incision opening to last incision closure
intraoperative bleeding | intraoperative
  Total amount of blood (mL) lost during the surgical procedure
postoperative drainage volume | two weeks after surgery
  Total amount of fluid (mL) collected through the chest drain during in-hospital stay
surgical mortality | 90 days after surgery
  Fatal complications occurryng within 90 days after surgery
complications | 30 days after surgery
  Any adverse event recorded perioperatively or after the surgical procedure during in-hospital stay
hospital stay | 30 days after surgery
  Overall duration (days) of in-hospital stay after the surgical procedure
a difference ≥10% in the score calculated for the exposure ergonomical domain. | one week after surgery
  3 ergonomical domains: exposure, instrumentation and maneuvering are assessed by 4 thoracic surgeons using a new scoring scale (score range 1, unsatisfactory to 3 excellent). Primary outcome is a difference ≥10% (sd=0.3) in at least one of the evaluated domains.
a difference ≥10% in the score calculated for the instrumentation ergonomical domain. | one week after surgery
  3 ergonomical domains: exposure, instrumentation and maneuvering are assessed by 4 thoracic surgeons using a new scoring scale (score range 1, unsatisfactory to 3 excellent). Primary outcome is a difference ≥10% (sd=0.3) in at least one of the evaluated domains.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Pompeo, MD, Principal Investigator — Tor Vergata University
Locations (1):
- Policlinico Tor Vergata University, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott WJ, Allen MS, Darling G, Meyers B, Decker PA, Putnam JB, McKenna RW, Landrenau RJ, Jones DR, Inculet RI, Malthaner RA. Video-assisted thoracic surgery versus open lobectomy for lung cancer: a secondary analysis of data from the American College of Surgeons Oncology Group Z0030 randomized clinical trial. J Thorac Cardiovasc Surg. 2010 Apr;139(4):976-81; discussion 981-3. doi: 10.1016/j.jtcvs.2009.11.059. Epub 2010 Feb 20. PMID 20172539
- [Background] Villamizar NR, Darrabie MD, Burfeind WR, Petersen RP, Onaitis MW, Toloza E, Harpole DH, D'Amico TA. Thoracoscopic lobectomy is associated with lower morbidity compared with thoracotomy. J Thorac Cardiovasc Surg. 2009 Aug;138(2):419-25. doi: 10.1016/j.jtcvs.2009.04.026. PMID 19619789
- [Background] Xu Y, Chen N, Ma A, Wang Z, Zhang Y, Liu C, Liu L. Three-dimensional versus two-dimensional video-assisted thoracic surgery for thoracic disease: a meta-analysis. Interact Cardiovasc Thorac Surg. 2017 Dec 1;25(6):862-871. doi: 10.1093/icvts/ivx219. PMID 29049786
- [Background] Bagan P, De Dominicis F, Hernigou J, Dakhil B, Zaimi R, Pricopi C, Le Pimpec Barthes F, Berna P. Complete thoracoscopic lobectomy for cancer: comparative study of three-dimensional high-definition with two-dimensional high-definition video systems dagger. Interact Cardiovasc Thorac Surg. 2015 Jun;20(6):820-3. doi: 10.1093/icvts/ivv031. Epub 2015 Mar 3. PMID 25736286
- [Background] Jiao P, Wu QJ, Sun YG, Ma C, Tian WX, Yu HB, Tong HF. Comparative study of three-dimensional versus two-dimensional video-assisted thoracoscopic two-port lobectomy. Thorac Cancer. 2017 Jan;8(1):3-7. doi: 10.1111/1759-7714.12387. Epub 2016 Oct 4. PMID 27755803
- [Background] Dong S, Yang XN, Zhong WZ, Nie Q, Liao RQ, Lin JT, Wu YL. Comparison of three-dimensional and two-dimensional visualization in video-assisted thoracoscopic lobectomy. Thorac Cancer. 2016 Sep;7(5):530-534. doi: 10.1111/1759-7714.12361. Epub 2016 May 23. PMID 27766782
- [Background] Yan TD, Black D, Bannon PG, McCaughan BC. Systematic review and meta-analysis of randomized and nonrandomized trials on safety and efficacy of video-assisted thoracic surgery lobectomy for early-stage non-small-cell lung cancer. J Clin Oncol. 2009 May 20;27(15):2553-62. doi: 10.1200/JCO.2008.18.2733. Epub 2009 Mar 16. PMID 19289625